CLINICAL TRIAL: NCT07220408
Title: A Single Center, Randomized, Double-masked, Vehicle Controlled Phase 2 Study Evaluating the Safety and Efficacy of TL-925 Ophthalmic Emulsion 0.1% Compared to Vehicle for the Treatment of Seasonal Allergic Conjunctivitis in the Conjunctival Allergen Challenge (Ora-CAC®) Model
Brief Title: Evaluation of TL-925 for the Treatment of Seasonal Allergic Conjunctivitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Telios Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TL-925-314
Record Dates: First submitted 2025-10-21; First posted 2025-10-23 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- TL-925 Arm (Active Comparator): Subjects will be dosed in clinic.
  Interventions: Drug: TL-925
- Placebo Arm (Placebo Comparator): Subjects wil be dosed in clinic.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TL-925 — TL-925 is an eye drop.
  Arms: TL-925 Arm
Drug: Placebo — The composition of the placebo is identical to the active formulation except for the exclusion of the active ingredient.
  Arms: Placebo Arm

SUMMARY:
In this prospective, Phase 2, randomized, double-masked, vehicle controlled study, approximately 60 eligible subjects will be randomized 1:1 to receive either TL-925 or placebo as topical ophthalmic eye drops administered bilaterally.

The study comprises of a screening and treatment period using the conjunctival allergen challenge model to evaluate TL-925 for the treatment of allergic conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 years or older
* Female subjects of childbearing potential and their male partners must both use a highly effective contraception method during the study.
* Documented history of ocular allergies and a positive skin test reaction to a seasonal (grass, ragweed, tree pollen) or perennial (cat dander, dog dander, dust mites, cockroach) allergen as confirmed by an allergic skin test conducted at Visit 1 or within the past 60 months.
* Calculated best-corrected visual activity
* Positive bilateral CAC reaction

Exclusion Criteria:

* Any systemic or ocular disease currently producing ocular redness and/or ocular discomfort, or that may interfere with the conduct of the study.
* Any ocular surgical intervention within the last 3 months OR refractive surgery within the last 6 months
* Any ongoing ocular infection (bacterial, viral or fungal)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-23 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Ocular Itching | 3, 5 and 7 minutes after CAC
  Ocular itching score will be reported by the subject at 3 timepoints after CAC at Visits 4d , 5d, and 6c.
Conjunctival Redness | 7, 15 and 20 minutes after CAC
  Conjunctival redness score will be evaluated by the investigator at 3 timepoints after CAC at Visits 4d, 5d, and 6c.

CONTACTS AND LOCATIONS:
Locations (1):
- Advancing Vision Research, Smyrna, Tennessee, United States